CLINICAL TRIAL: NCT05963477
Title: Pediatric Post-operative Abdominal Wound Dehiscence in Association With Midline vs Other Incisions in Tertiary Care Setting Kabul Afghanistan: A Cohort Study
Brief Title: Pediatric Post-operative Abdominal Wound Dehiscence in Association With Midline vs Other Incisions: A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: French Medical Institute for Mothers and Children (Other Government)
Responsible Party: Principal Investigator, Abdullah Bahloli, Dr. Abdullah Bahloli, French Medical Institute for Mothers and Children
Other Study IDs: 40-FMIC-ER-18
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Wound Dehiscence; Incision
Keywords: abdominal wound dehiscence, burst abdomen, pediatric abdominal incisions, children
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Age Group: Neonates Infants Children
  Interventions: Procedure: laparatomy
- Gender: Male Female
  Interventions: Procedure: laparatomy
- Selective/Emergency: Selective Emergency
  Interventions: Procedure: laparatomy
- Wound Class: Clean Clean-contaminated Contaminated Infected
  Interventions: Procedure: laparatomy
- Risk Factors: Yes No
  Interventions: Procedure: laparatomy
- Type of Incisions: Midline Trransverse Oblique
  Interventions: Procedure: laparatomy

INTERVENTIONS:
Procedure: laparatomy — all abdominal procedures which are approached by different incisions

SUMMARY:
This study is designed to see different abdominal incisions complication among neonates, infants and children and to find risk factors for developing wound dehiscence

ELIGIBILITY:
Inclusion Criteria:

-all abdominal surgeries patient under 18-year-old.

Exclusion Criteria:

* Umbilical hernia, redo laparatomy, laparoscopic surgery.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all patients from neonatal age until 18 years old who were planned to undergo abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Wound dehiscence or burst abdomen | one month after intervention
  the overall outcome of the intervention (incisions) is wound dehiscence in different age groups, in gender, among who has or has no risk factors and among different wound class

CONTACTS AND LOCATIONS:
Locations (1):
- French Medical Institute for Mothers and Children, Kabul, Afghanistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT05963477/Prot_SAP_000.pdf